CLINICAL TRIAL: NCT05806736
Title: Study on the Efficacy and Mechanism of Transcutaneous Auricular Vagus Nerve Stimulation in the Treatment of Sleep Disorders in Parkinson's Disease
Brief Title: Curative Effect and Mechanism of Transcutaneous Auricular Vagus Nerve Stimulation on Sleep Disorders of PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kezhong Zhang, professor/Chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-SR-519
Record Dates: First submitted 2023-02-27; First posted 2023-04-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: non-motor symptoms; Therapeutics; nighttime insomnia
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active transcutaneous auricular vagus nerve stimulatio (Experimental): For Experimental Arm, active transcutaneous auricular vagus nerve stimulation, Patients underwent fourteen consecutive daily sessions of taVNS.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation (real stimulation)
- sham transcutaneous auricular vagus nerve stimulation (Sham Comparator): For sham transcutaneous auricular vagus nerve stimulation arm, Sham Comparator, patients underwent fourteen consecutive daily sessions of sham-taVNS (the electrodes were fixed at the left earlobe with the same stimulation parameters).
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation (sham stimulation)

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation (real stimulation) — Transcutaneous auricular vagus nerve stimulation was conducted by transcutaneous electrical stimulation therapy instrument to the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve. Stimulation parameters: frequency = 20/4 Hz; pulse width = 200 μs, twice a day, 30 minutes each time.
  Arms: active transcutaneous auricular vagus nerve stimulatio
Device: Transcutaneous auricular vagus nerve stimulation (sham stimulation) — Transcutaneous auricular vagus nerve stimulation was conducted by transcutaneous electrical stimulation therapy instrument to the left earlobe. Stimulation parameters: frequency = 20/4 Hz; pulse width = 200 μs, twice a day, 30 minutes each time.
  Arms: sham transcutaneous auricular vagus nerve stimulation

SUMMARY:
This study is a double-blind comparative study examining the curative effect and mechanism of the transcutaneous auricular vagus nerve stimulation treatment on non-motor symptoms of Parkinson's disease patients. The investigators hypothesize that treatment using transcutaneous auricular vagus nerve stimulation will improve the non-motor symptoms, such as improving sleep, and improve cortical activity simultaneously in Parkinson's disease patients.

DETAILED DESCRIPTION:
Patients in the Experimental group underwent fourteen consecutive daily sessions of transcutaneous auricular vagus nerve stimulation (taVNS, twice daily, 30 minutes each time), whereas patients in the sham stimulation group underwent fourteen consecutive daily sessions of sham taVNS. Assessments of motor and non-motor symptoms, cortical activity (using Functional near-infrared spectroscopy) and blood indicators were performed three times: at baseline, one day post intervention, fourteen days post intervention.

ELIGIBILITY:
Inclusion Criteria:

(i) right-handed individuals aged 45-80 years; (ii) met the diagnostic criteria for idiopathic PD and had been stable on medication for at least one month; (iii) met the diagnostic criteria for insomnia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, and insomnia had to have lasted for at least six months, with Pittsburgh sleep quality index (PSQI) scores >7; (iv) no history of medication that might affect the study, such as sleeping pills or antidepressants, that is, the PSQI hypnotic medication score of 0; (v) clear consciousness, basic communication skills and cooperation in all assessments and treatments; (vi) The patients agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

(i) those with concomitant cognitive dysfunction, such as Montreal cognitive assessment (MoCA) <23; (ii) those with secondary Parkinson's syndrome or Parkinson's superimposed syndrome; (iii) those with severe cardiac, pulmonary, hepatic, renal, or concomitant malignancies or a history of previous brain surgery; (iv) those with contraindications to taVNS interventions; (v) those with severe psychiatric disorders; (vi) Insomnia not caused by PD, such as frequent (two times per week) nighttime use of sedative medications (including sedative antidepressants), untreated restless legs syndrome, night-shift work or other occupations that result in abnormal sleep patterns, insomnia associated with dopamine therapy, and other reversible causes of insomnia identified by the baseline clinical interview.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in sleep quality, sleep efficiency of patients | Assessed at baseline, one day post intervention, fourteen days post intervention.
  Pittsburgh sleep quality index (PSQI) was used to evaluate the sleep quality of participants in the past month. It consists of 19 self-evaluation and 5 other evaluation items. The total score range is 0-21, with higher scores indicating poorer sleep quality.

SECONDARY OUTCOMES:
The motor part of the Unified Parkinson's Disease Rating Scale | Assessed at baseline, one day post intervention, fourteen days post intervention.
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms. The minimum and maximum values of the motor part of the Unified Parkinson's Disease Rating Scale are 0 and 108. A higher score means a worse outcome.
Changes of sleep quality scale | Assessed at baseline, one day post intervention, fourteen days post intervention.
  Non-motor symptoms such as sleep disorders were evaluated by Parkinson's disease sleep scale-2 (PDSS-2). PDSS-2 is an improved version of PDSS used to screen for common types of sleep disorders in Parkinson's disease patients. The minimum and maximum values of the non-motor part of the PDSS-2 Scale are 0 and 60. A higher score means a worse outcome.
Changes of Rapid-eye-movement Sleep Behavior Disorder scale | Assessed at baseline, one day post intervention, fourteen days post intervention.
  Rapid-eye-movement Sleep Behavior Disorder Screening Questionnaire (RBDSQ) was used to assess the behavior disorder of multiple eye movement sleep. The minimum and maximum values of the non-motor part of the RBDSQ Scale are 0 and 13. A higher score means a worse outcome.
Epworth sleepiness scale (ESS) | Assessed at baseline, one day post intervention.
  The Epworth Sleepiness Scale, also known as the Epworth Daytime Sleepiness Scale, was developed by Johns MW to assess excessive daytime sleepiness. This scale has clinical significance: it can provide a semi-objective assessment of sleepiness. Scoring more than 6 out of 24 indicates drowsiness, more than 11 indicates excessive sleepiness, and more than 16 indicates dangerous sleepiness.
Hamilton Depression Scale-24 (HAMD-24) | Assessed at baseline, one day post intervention.
  The Hamilton Depression Rating Scale is the most widely used instrument for clinical assessment of depressive states, effectively reflecting the severity of the condition. The total score ranges from 0 to 76 points, with lower scores indicating milder symptoms and higher scores signifying more severe conditions.
Hamilton Anxiety Scale (HAMA) | Assessed at baseline, one day post intervention.
  The Hamilton Anxiety Scale is commonly used in clinical practice as a basis for diagnosing anxiety disorders and assessing their severity. The total score can be used to evaluate the severity of anxiety symptoms in patients with anxiety and depressive disorders, as well as to assess the effects of various pharmacological and psychological interventions. According to data provided by the Chinese Scale Collaborative Group: a total score ≥29 indicates possible severe anxiety; ≥21 confirms significant anxiety; ≥14 confirms the presence of anxiety; >7 suggests possible anxiety; and a score <7 indicates no anxiety symptoms.
Montreal Cognitive Assessment (MoCA) | Assessed at baseline, one day post intervention.
  The Montreal Cognitive Assessment is an evaluation tool used for rapid screening of patients with mild cognitive impairment. The assessed cognitive domains include attention and concentration, executive function, memory, language, visuospatial skills, abstract thinking, as well as calculation and orientation. The total score of the scale is 30 points, with test results indicating a normal value of ≥26 points.
Changes in ΔHbO2 concentration in the brain cortex | Assessed at baseline, one day post intervention.
  The ΔHbO2 concentration in the brain cortex will be recorded in oxyhemoglobin.
Plasma indicators | Assessed at baseline, one day post intervention, fourteen days post intervention.
  5ml of the patient's elbow vein blood was collected and centrifuged after standing and stratified. The blood plasma was collected and frozen at - 20 ℃ for testing. Detection of changes in plasma ghrelin levels.
Subjective sleep assessment | Assessed at baseline, one day post intervention, fourteen days post
  Using sleep logs to record participants' subjective sleep data, including subjective sleep quality scores，early morning refreshment scores, easy wake up scores, ease of falling asleep scores, and dreaming scores.
Objective sleep assessment | Assessed at baseline, one day post intervention, fourteen days post
  Using MI wristbands for objective sleep assessment, including deep sleep time scores，night waking up times, light sleep duration, and the REM sleep duration.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No